CLINICAL TRIAL: NCT04623502
Title: An Investigation of Kidney and Urothelial Tumor Metabolism in Patients Undergoing Surgical Resection and/or Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Howard Hughes Medical Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vitaly Margulis, Principal Investigator, Professor of Urology, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2019-1061; P50CA196516 (NIH); R35CA220449 (NIH); F31CA239330 (NIH); HHMI Investigator:DeBerardinis (Other Grant/Funding Number: Howard Hughes Medical Institute)
Record Dates: First submitted 2020-10-19; First posted 2020-11-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma; Clear Cell Carcinoma; Urothelial Carcinoma; Metastatic Kidney Cancer; Metastatic Urothelial Carcinoma; Papillary Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Fumarate Hydratase Deficiency; Succinate Dehydrogenase-Deficient Renal Cell Carcinoma; HLRCC; Hereditary Leiomyomatosis and Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Adenocarcinoma, Clear Cell; Carcinoma, Transitional Cell; Fumaric aciduria; Hereditary leiomyomatosis and renal cell cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 13C-Glucose (Experimental)
  Interventions: Other: 13C-Glucose
- 13C-Acetate (Experimental)
  Interventions: Other: 13C-Acetate
- 13C-Lactate (Experimental)
  Interventions: Other: 13C-Lactate
- 13C-Glutamine (Experimental)
  Interventions: Other: 13C-Glutamine
- 13C-Fructose (Experimental)
  Interventions: Other: 13C-Fructose

INTERVENTIONS:
Other: 13C-Glucose — Patients in the 13C-glucose arm will receive an infusion of a 13C-glucose solution. In most cases, the glucose infusion will be administered for 2-3 hours prior to resection of the mass. During the surgical procedure, 2-4mL of blood will be obtained approximately every 30 minutes to monitor blood glucose and/or blood pH. The infusion will be stopped after resection.
  Arms: 13C-Glucose
Other: 13C-Acetate — Patients in the 13C-acetate arm will receive an infusion of a 13C-acetate solution. In most cases, the acetate infusion will be administered for 2-3 hours prior to resection of the mass. During the surgical procedure, 2-4mL of blood will be obtained approximately every 30 minutes to monitor blood glucose and/or blood pH. The infusion will be stopped after resection.
  Arms: 13C-Acetate
Other: 13C-Lactate — Patients in the 13C-lactate arm will receive an infusion of a 13C-lactate solution. In most cases, the lactate infusion will be administered for 2-3 hours prior to resection of the mass. During the surgical procedure, 2-4mL of blood will be obtained approximately every 30 minutes to monitor blood glucose and/or blood pH. The infusion will be stopped after resection.
  Arms: 13C-Lactate
Other: 13C-Glutamine — Patients in the 13C-glutamine arm will receive an infusion of a 13C-glutamine solution. In most cases, the glutamine infusion will be administered for 2-3 hours prior to resection of the mass. During the surgical procedure, 2-4mL of blood will be obtained approximately every 30 minutes to monitor blood glucose and/or blood pH. The infusion will be stopped after resection.
  Arms: 13C-Glutamine
Other: 13C-Fructose — Patients in the 13C-fructose arm will receive an infusion of a 13C-fructose solution. In most cases, the fructose infusion will be administered for 2-3 hours prior to resection of the mass. During the surgical procedure, 2-4mL of blood will be obtained approximately every 30 minutes to monitor blood glucose and/or blood pH. The infusion will be stopped after resection.
  Arms: 13C-Fructose

SUMMARY:
The purpose of this study is to understand the metabolism of cancers involving the kidney, including renal cell carcinomas and urothelial cell carcinomas, and how kidney cancers use different types of fuel to support tumor growth. This study uses specially labeled nutrient tracers of compounds normally found circulating in the blood. The nutrients (glucose, fructose, glutamine, acetate, and lactate) are also found in common foods. A nutrient tracer will be given to the participants through an intravenous (IV) catheter during surgery or biopsy, and blood will be collected every 30 minutes during the infusion to monitor safety parameters and the nutrient tracers. The investigators will collect a tissue sample after the completion of surgery. Participants not having an infusion will have their tissue collected after surgery or biopsy.

Participation in this study will not change patient care. All patients will receive standard of care treatment as determined by their doctors.

DETAILED DESCRIPTION:
The purpose of this study is to understand the metabolism of kidney cancers (renal cell carcinomas and urothelial cell carcinomas involving the kidney) in patients. Metabolism is the term used to describe how cells take up different nutrients and convert them to energy and materials needed for cell growth. In cancer, metabolism is hijacked to support the needs of cancer cells. Cancer cells can use multiple nutrients in the blood to fuel their growth, but it is not known what materials cancer cells make with those nutrients in patients.

Many participants in this study will be infused with a 13C-labeled nutrient during their surgery or biopsy. 13C means that the carbon in the nutrient is heavier than 12C carbons that are the most abundant carbon atoms in nature. 13C carbons account for about 1% of natural carbon atoms are not radioactive or harmful in any way. Using the tissue collected during or after surgery and/or biopsy, the researchers can track how the heavier 13C carbons from the infused nutrient are being used to make different materials that cancer cells need to grow.

The researchers hope to understand how kidney cancers change their metabolism to adapt, grow, and survive in patients. The knowledge learned from this study will be used to support the development of therapies that target metabolic adaptations, and the development of new non-invasive imaging techniques that will improve the care and survival of future kidney cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic evidence of known or probable kidney or urothelial cancer requiring surgical biopsy or excision.
* Age ≥ 18 years
* Subjects of all races and ethnic origins
* The willingness to sign and ability to understand a written informed consent.
* Patients participating in other clinical trials are eligible, and will be evaluated on a case by case basis by the Principal Investigator, Dr. Vitaly Margulis, MD.

Exclusion Criteria:

* Uncontrolled or poorly controlled diabetes for patients receiving a 13C infusion
* Pregnant or breastfeeding
* Not a surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent of 13C isotopologue distributions | 5 years
  Tissue and blood samples will be analyzed for 13C isotopologue distributions (percent) in central carbon metabolites using mass spectrometry. This allows the Investigators to understand how different subtypes of kidney and urothelial cancers alter utilization of the 13C tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Margulis, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States